CLINICAL TRIAL: NCT05938517
Title: Pharmacokinetic Profile of Betahistine Serum Concentration With and Without Selegiline in Healthy Volunteers - a Prospective Mono-center Open-labeled Phase I Trial ("PK-BeST")
Brief Title: Pharmacokinetic Profile of Betahistine With and Without Selegiline in Healthy Volunteers
Acronym: PK-BesT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Michael Strupp, Senior physician, Ludwig-Maximilians - University of Munich
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19-0992 fed
Record Dates: First submitted 2023-06-26; First posted 2023-07-10 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Ménière's Disease
Keywords: Betahistine-dihydrochloride; Selegiline-hydrochloride; MAO-B inhibitor
MeSH Terms: conditions — Meniere Disease | interventions — Betahistine; Selegiline

STUDY DESIGN:
Intervention Model Description: Subjects satisfying all selection criteria were included in the open-labeled trial receiving 3 different dosages of Betahistine alone in ascending order (24 mg, 48 mg, 96 mg) in the first period. In the second period, subjects received Betahistine treatment as described for first period but after pre- and continuous treatment with 5 mg/ml Selegiline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Betahistine-dihydrochloride (Experimental): Subjects received single dosages of Betahistine (24 mg, 48 mg, 96 mg) orally for pharmacokinetic serum draw with at least two days between the different dosages.
  Interventions: Drug: Betahistine dihydrochloride
- Betahistine-dihydrochloride and Selegiline-hydrochloride (Experimental): Subjects were pre-treated with Selegiline (5 mg/day) orally for one week and treated continuously with Selegiline (5 mg/day) in combination with the single dosages of Betahistine (24 mg, 48 mg, 96 mg) orally with at least two days between the different dosages.
  Interventions: Drug: Betahistine dihydrochloride; Drug: Selegiline-hydrochloride

INTERVENTIONS:
Drug: Betahistine dihydrochloride — Each subject received single dosages of Betahistine (24 mg, 48 mg, 96 mg) for pharmacokinetic serum draw with at least two days between the different dosages.
  Other Names: Vasomotal
Drug: Selegiline-hydrochloride — In the second period, each subject was pre-treated with Selegiline (5 mg/day) for one week and treated continuously with Selegiline (5 mg/day) in combination with the single dosages of Betahistine (24 mg, 48 mg, 96 mg) with at least two days between the different dosages.
  Other Names: Selegiline-neuraxpharm
  Arms: Betahistine-dihydrochloride and Selegiline-hydrochloride

SUMMARY:
The goal of this pharmakokinetic trial is to demonstrate that Betahistine serum concentration is higher after combination treatment with Betahistine and Selegiline compared to Betahistine alone.

The main questions it aims to answer are:

Is the plasma concentration of betahistine higher due to combination treatment with selegiline compared to betahistine monotherapy? How is the safety of the combination treatment with betahistine and selegiline, the pharmacokinetics of betahistine in different dosages in blood, and the inter-individual differences in the metabolism?

Subjects satisfying all selection criteria will receive three different dosages of Betahistine alone orally in ascending order (24 mg, 48 mg, 96 mg) in the first period. In the second period, subjects received Betahistine treatment as described for first period but after pre- and continuous treatment with 5 mg/ml Selegiline orally. Plasma concentration (namely the AUC0-240min) of betahistine will be measured before and 10, 30, 60, 90, 120, 180, 240 minutes after treatment with blood examinations. Safety parameters include assessment of adverse events, ECG, vital signs, laboratory measurements including kidney and liver function, full blood count and pregnancy and drug screening test.

DETAILED DESCRIPTION:
This study was an investigator-initiated (IIT) prospective mono-center open-labeled trial to demonstrate that Betahistine serum concentration is higher after combination treatment with Betahistine and Selegiline compared to Betahistine alone in healthy subjects.

Subjects were screened for their eligibility to participate in the study. Each subject gave written informed consent before any study-related procedures were performed.

Subjects satisfying all selection criteria were included in the open-labeled trial receiving 3 different dosages of Betahistine alone in ascending order (24 mg, 48 mg, 96 mg) in the first period. In the second period, subjects received Betahistine treatment as described for first period but after pre- and continuous treatment with 5 mg/ml Selegiline. Betahistine serum concentrations were measured over a period of 240 min at 8 time points (area under the curve, AUC0-240 min). Safety parameters included assessment of adverse events, ECG, vital signs, laboratory measurements including kidney and liver function, full blood count and pregnancy and drug screening test). Safety monitoring was conducted during every visit and assessment of vital parameter and adverse events were conducted 10, 30, 60, 90, 120, 180, and 240min after betahistine intake. The clinical trial was conducted in a hospital of maximum care with the possibility to consult a specialist for possible symptoms of an intoxication especially an anesthesiologist, cardiologist and neurologist 24 hours/7 days a week.

ELIGIBILITY:
Diagnosis and main criteria for inclusion:

* Adult healthy volunteers, males and non-pregnant, non-breastfeeding woman with adequate contraception
* Subjects must meet all of the following inclusion criteria to be eligible for enrolment into the trial:
* Healthy volunteers (age ≥ 18 years and ≤ 70 years) as determined by screening
* and Principal Investigator's judgement
* No intake of medication due to an illness
* Written informed consent of the subject
* Systolic blood pressure between 90 and 140 mmHg and diastolic blood pressure between 60 and 90 mmHg at screening
* PQ interval in the ECG between 0.12 s and 0.20 s
* Duration of the QRS complex between 0.06 s and 0.10 s
* QTc interval 440 ms or less
* Heart rate between 60 and 100 beats per minute
* Subjects with the ability to follow study instructions and likely to attend and complete all required visits

Subjects presenting with any of the following exclusion criteria were not included in the trial:

* Subject is not able to give consent
* A condition in which repeated serum draws or injections pose more than minimal risk for the subjects, such as haemophilia, other severe coagulation disorders or significantly impaired venous access
* Participation in another study with an investigational drug or device within the last 30 days, prior participation in the present study, or planned participation in another trial
* Intake of medication due to an illness
* Subjects with a physical or psychiatric condition which at the investigator's discretion may put the subject at risk, may confound the trial results, or may interfere with the subject's participation in the clinical trial before participation in this study
* Current or planned pregnancy or breastfeeding woman
* Woman of childbearing potential who is not willing to use medically reliable methods of contraception for the entire study duration
* Intake of alcohol 24 hours before first IMP intake or during study participation
* Known or persistent abuse of medication, drugs or alcohol (positive test for alcohol or drugs)
* Known contraindications for Betahistine, such as bronchial asthma, pheochromocytoma, treatment with antihistaminic drugs, ulcer of the stomach or duodenum, severe dysfunction of liver or kidney, hypersensitivity to Betahistine or other ingredients
* Known contraindications for Selegiline, e.g. use of opioids, tricyclic antidepressants, sympathomimetics, non-selective MAOIs, (selective) serotonin (-noradrenaline) re-uptake inhibitors (SSRI/SNRI), serotonin agonists, hypersensitivity to Selegiline or other ingredients
* Hereditary intolerance to galactose, hereditary deficiency of lactose, glucose-galactose-malabsorption
* AV Block in the ECG
* Hypotonic or hypertonic subjects according to the criteria of the National Heart, Lung and Serum Institute (Hypertension > 90/140 mmHg, Hypotension < 90/60 mmHg)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Mean AUC of Betahistine | 240 minutes
  Mean AUC of Betahistine in serum after treatment of Betahistine alone or with Selegiline

SECONDARY OUTCOMES:
Mean Half Life of Betahistine | 240 minutes
  Half Life of Betahistine following the administration of different Betahistine doses with and without Selegiline
Occurrence of adverse effects | up to 8 weeks
  Occurrence of adverse effects following the administration of different Betahistine doses with and without Selegiline

CONTACTS AND LOCATIONS:
Overall Officials: Michael Strupp, M.D., Principal Investigator — LMU Munich
Locations (1):
- Department of Neurology, Ludwig Maximilian University, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strupp M, Churchill GC, Naumann I, Mansmann U, Al Tawil A, Golentsova A, Goldschagg N. Examination of betahistine bioavailability in combination with the monoamine oxidase B inhibitor, selegiline, in humans-a non-randomized, single-sequence, two-period titration, open label single-center phase 1 study (PK-BeST). Front Neurol. 2023 Oct 18;14:1271640. doi: 10.3389/fneur.2023.1271640. eCollection 2023. PMID 37920833